CLINICAL TRIAL: NCT05049239
Title: Support in Activity, Movement and Exercise-for Adults with ADHD. a Randomized Controlled Trial Intervention Study with 12 Weeks of Physical Training with and Without Cognitive Support.
Brief Title: Structured Physical Training with and Without Cognitive Support for Adults with ADHD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OLL-274569
Record Dates: First submitted 2021-05-14; First posted 2021-09-20 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: ADHD
Keywords: Physical exercise; Cognitive support; Group intervention
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Motor Activity | interventions — Physical Conditioning, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Physical training (Experimental): Medium-high-intensity physical training 3 times a week, 60 min / time for 12 weeks.
  Interventions: Behavioral: Physical training
- Physical training combined with cognitive support (Active Comparator): Medium-high-intensity physical training 3 times a week, 60 min / time for 12 weeks.
  The cognitive support consists of person centred individual occupational therapy.
  Interventions: Behavioral: Physical training combined with cognitive support.
- Control group (No Intervention): The control group receive no intervention.

INTERVENTIONS:
Behavioral: Physical training — Medium-high-intensity physical training 3 times a week, 60 min / time for 12 weeks, consisting of fitness, strength and mobility exercises with a target level of 60-90% of maximum heart rate. Two sessions per week take place in a group led by a physiotherapist and once a week the training consists of self-chosen training individually or in group.
  Arms: Physical training
Behavioral: Physical training combined with cognitive support. — Medium-high-intensity physical training 3 times a week, 60 min / time for 12 weeks, consisting of fitness, strength and mobility exercises with a target level of 60-90% of maximum heart rate. Two sessions per week take place in a group led by a physiotherapist and once a week the training consists of self-chosen training individually or in group.
  The cognitive support consists of person centred individual occupational therapy with focus on daily time management skills and planning and organisation in daily life, i.e. make time for physical exercise. The number of session during the intervention period depend on the participants needs and is estimated to 4-6 sessions.
  Arms: Physical training combined with cognitive support

SUMMARY:
Studies in children and adolescents with Attention-Deficit-Hyperactivity-Disorder (ADHD) have shown that physical exercise can improve the core symptoms of ADHD; inattention and hyperactivity. For adults, the evidence is deficient and there is a great need to investigate whether adults have the same effect on ADHD symptoms of physical exercise, as children and young people have. Adults with ADHD often have a sedentary lifestyle and suffer from obesity and have sleep problems. In a normal population, these problems have been shown to be affectable with physical exercise. START (Support in Activity, Movement and Exercise) is a randomized controlled intervention study where physical exercise is given for 12 weeks, with or without cognitive support. The effect is measured with rating scales as well as cognitive and physical tests. The purpose is to investigate whether START works as a treatment for ADHD in terms of ADHD symptoms and disability, and what impact the intervention has on mental health, physical condition and activity level, body awareness and everyday functioning.

Outcome measures are registered within 3 weeks before and after the end of treatment, after 6 months and 12 months. The randomization takes place in three groups; physical exercise (i), physical exercise and extra cognitive support (ii), and control group on waiting list (iii).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ADHD.

Exclusion Criteria:

* Ongoing depression with points on MADRS-S over 21
* Suicidality
* Bipolar disorder
* Psychosis
* Ongoing addiction
* Reported threatening behavior.
* Severe autism that makes group participation impossible
* Inability to read and understand the Swedish language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Clinical Global Impression-Improvement (CGI-I) | Pre-intervention, post-intervention (12 weeks) and 3, 6 and 12 months after intervention start
  Assess total improvement on a Richter scale. Range 1-7, Higher scores mean worse outcome
Changes in Adult ADHD Self-Report Scale (ASRS-v.1.1) | Pre-intervention, post-intervention (12 weeks) and 3, 6 and 12 months after intervention start
  Range 0-72, higher scores mean worse outcome

SECONDARY OUTCOMES:
Changes in Cardio Respiratory Fitness | Pre-intervention, post-intervention (12 weeks) and 3, 6 and 12 months after intervention start
  Measured in millilitre per kilogram per minute with the Ekblom-Bak test, a submaximal exercise test.
  Higher value means better outcome
Changes in Balance | Pre-intervention, post-intervention (12 weeks) and 3, 6 and 12 months after intervention start
  Measured with Flamingo test. The test person is standing on the preferred leg on a low balance profile for 60 seconds. The number of times that the test person puts his/her foot to the ground is counted. Lower value means better outcome
Changes in Body Mass Index | Pre-intervention, post-intervention (12 weeks) and 3, 6 and 12 months after intervention start
  Weight and height will be measured in kilograms and centimeters, and combined to report BMI in kg/m^2.
  Lower value means better outcome
Changes in Abdominal Circumference | Pre-intervention, post-intervention (12 weeks) and 3, 6 and 12 months after intervention start
  Measured with a measuring tape in centimeters. Lower value means better outcome
Changes in Body Awareness | Pre-intervention, post-intervention (12 weeks) and 3, 6 and 12 months after intervention start
  Body Awareness Scale - movement quality and experience (BAS MQ-E). Higher value means better outcome.
Changes in Blood pressure | Pre-intervention, post-intervention (12 weeks) and 3, 6 and 12 months after intervention start
  Both systolic and diastolic blood pressure will be measured in mm Hg with a blood pressure monitor on the arm.
Changes in Satisfaction with Daily Occupations-Occupational Balance (SDO-OB) activity score | Pre-intervention, post-intervention (12 weeks) and 3, 6 and 12 months after intervention start
  Range 0-17, higher scores are better
Changes in Satisfaction with daily occupations and occupational balance (SDO-OB) satisfaction score | Pre-intervention, post-intervention (12 weeks) and 3, 6 and 12 months after intervention start
  Global satisfaction score, range 1-5, lower scores are better
Changes in Canadian Occupational Performance Measure (COPM) perfomance score | Pre-intervention, post-intervention (12 weeks) and 3, 6 and 12 months after intervention start
  Range 5-50, higher scores are better
Changes in Canadian Occupational Performance Measure (COPM) satisfaction score | Pre-intervention, post-intervention (12 weeks) and 3, 6 and 12 months after intervention start
  Range 5-50, higher scores are better
Changes in Adult ADHD Quality of Life Measure (AAQoL) | Pre-intervention, post-intervention (12 weeks) and 3, 6 and 12 months after intervention start
  Range 29-145, higher scores are better
Changes in Self Efficacy Scale (GSE-10) | Pre-intervention, post-intervention (12 weeks) and 3, 6 and 12 months after intervention start
  Range 0-40, higher scores are better
Changes in Assessment of Time Management Skills-Swedish (ATMS-S) Time management subscale | Pre-intervention, post-intervention (12 weeks) and 3, 6 and 12 months after intervention start
  11 items, reported as 0-100 ATMS units, higher scores are better
Changes in Assessment of Time Management Skills-Swedish (ATMS-S), Organization and planning sub scale | Pre-intervention, post-intervention (12 weeks) and 3, 6 and 12 months after intervention start
  11 items, reported as 0-100 ATMS units, higher scores are better
Change in Assessment of Time Management Skills-Swedish (ATMS-S), Regulation of emotions sub scale | Pre-intervention, post-intervention (12 weeks) and 3, 6 and 12 months after intervention start
  5 items, reported as 0-100 ATMS units, higher scores are better
Changes in EuroQuality of Life - 5 dimensions - 5 levels (EQ-5D-5L): item scores | Pre-intervention, post-intervention (12 weeks) and 3, 6 and 12 months after intervention start
  5 items scored 1-5
Change in EuroQuality of Life - 5 dimensions - 5 levels (EQ-5D-5L): global score | Pre-intervention, post-intervention (12 weeks) and 3, 6 and 12 months after intervention start
  One visual-analogue-scale answer (range 0-100), higher scores are better
Changes in Continuous Performance Test (AX-CPT) | Pre-intervention, post-intervention (12 weeks) and 3, 6 and 12 months after intervention start
  Measures cognitive flexibility. Will be done in conjunction with functional Magnetic resonance imaging (fMRI).
Changes in GO/NoGO | Pre-intervention, post-intervention (12 weeks) and 3, 6 and 12 months after intervention start
  Measures impulse control. Will be done in conjunction with functional Magnetic resonance Imaging (fMRI)
Changes Affective Picture series (IAPS) | Pre-intervention, post-intervention (12 weeks) and 3, 6 and 12 months after intervention start
  Measures emotion regulation. Will be done in conjunction with functional Magnetic resonance imaging (fMRI)

OTHER OUTCOMES:
Changes in Cortical thickness | Pre-intervention, post-intervention (12 weeks) and 3, 6 and 12 months after intervention start
  Structural Magnetic resonance imaging (MRI)

CONTACTS AND LOCATIONS:
Overall Officials: Mussie Msghina, Assoc.Prof, Principal Investigator — Örebro University and Regional Örebro County
Locations (1):
- Öppenvårdspsykiatrisk mottagning, Universitetssjukhuset Örebro, Örebro, Örebro County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with researchers within the research group only.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will become available from study start to the end of the study
Access Criteria: To get access the person have to be involved in all parts of the study. Access is decided by PI. Access to data is password protected in accordance with the European General Data Protection Regulation (GDPR).

REFERENCES:
- [Derived] Svedell LA, Lindvall MA, Holmqvist KL, Cao Y, Msghina M. Physical exercise as add-on treatment in adults with ADHD - the START study: a randomized controlled trial. Front Psychiatry. 2025 Oct 30;16:1690216. doi: 10.3389/fpsyt.2025.1690216. eCollection 2025. PMID 41244864
- [Derived] Lindvall MA, Holmqvist KL, Svedell LA, Philipson A, Cao Y, Msghina M. START - physical exercise and person-centred cognitive skills training as treatment for adult ADHD: protocol for a randomized controlled trial. BMC Psychiatry. 2023 Sep 25;23(1):697. doi: 10.1186/s12888-023-05181-1. PMID 37749523
- [Derived] Svedell LA, Holmqvist KL, Lindvall MA, Cao Y, Msghina M. Feasibility and tolerability of moderate intensity regular physical exercise as treatment for core symptoms of attention deficit hyperactivity disorder: a randomized pilot study. Front Sports Act Living. 2023 May 15;5:1133256. doi: 10.3389/fspor.2023.1133256. eCollection 2023. PMID 37255729